CLINICAL TRIAL: NCT04091087
Title: A Phase 2, Randomized, Double-Blind, Vehicle-Controlled, Proof-of-Concept Study to Evaluate the Efficacy, Safety, and Local Tolerability of Crisaborole Ointment, 2%, in Adult Participants With Stasis Dermatitis Without Active Skin Ulceration
Brief Title: Study Evaluating Efficacy and Safety of Crisaborole in Adults With Stasis Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C3291038
Record Dates: First submitted 2019-09-13; First posted 2019-09-16 (Actual); Results first posted 2022-05-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Stasis Dermatitis
Keywords: Stasis Dermatitis; venous hypertension; venous insufficiency
MeSH Terms: conditions — Venous Insufficiency | interventions — crisaborole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- crisaborole ointment (Experimental): crisaborole ointment
  Interventions: Drug: crisaborole ointment
- vehicle ointment (Sham Comparator): vehicle ointment
  Interventions: Other: vehicle ointment

INTERVENTIONS:
Drug: crisaborole ointment — crisaborole ointment
  Other Names: Eucrisa
  Arms: crisaborole ointment
Other: vehicle ointment — vehicle ointment
  Arms: vehicle ointment

SUMMARY:
This is a Phase 2a, randomized, double blind, vehicle controlled, parallel group, proof of concept study that will include participants with stasis dermatitis without active skin ulceration, who will receive crisaborole ointment 2% or vehicle twice daily for 6 weeks.

DETAILED DESCRIPTION:
Study C3291038 is a Phase 2a, randomized, double-blind, vehicle-controlled, parallel-group, proof of concept study to evaluate the efficacy, safety, and local tolerability of 6 weeks of treatment with crisaborole in adult participants with SD without active skin ulceration. Approximately 70 eligible participants will be randomized into the double blind treatment period in a 1:1 ratio to receive crisaborole ointment, 2% or vehicle twice daily for 6 weeks.

The study will recruit male and female participants aged ≥ 45 years with a clinical diagnosis of SD.

The total duration of participation in the study will be up to 14 weeks, including up to 4 weeks for screening, a 6 week double blind treatment period, and a follow-up period of 4 weeks after treatment completion.

Study enrollment and management will be de centralized, where participants do not visit an investigator or a clinic for clinical assessment. The participants will participate in the study at home. The sponsor (or designee) will provide home visits by qualified home visit practitioners (HVP), remote contact by telemedicine (or telephone), and clinical database electronic case report forms (eCRFs), eDiary, and other electronic data entries from 3rd party vendors for study data collection.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are ≥45 years of age and in generally stable health
* Participants who are in generally stable health and have a known diagnosis of Stasis Dermatitis or newly diagnosed Stasis Dermatitis
* Participants whose mental and physical status allows them to be able to mostly perform their activities of daily living with minimal assistance

Exclusion Criteria:

* Participants with clinically significant active or potentially recurrent dermatitis conditions and known genetic dermatological conditions that are not Stasis Dermatitis or overlap with Stasis Dermatitis
* Participants with active venous stasis ulceration on either lower extremity.
* Participants with current infection or suspected infection of any Stasis Dermatitis lesions
* Women of child bearing potential (WOCBP) are not eligible for this study

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2020-06-26 (Actual); Primary Completion 2021-10-19 (Actual); Study Completion 2021-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (4):
  - Lightship, El Segundo, California
  - Hawthorne Effect, Inc, Lafayette, California
  - Verily Life Sciences LLC, South San Francisco, California
  - Onco360 Oncology Pharmacy, Louisville, Kentucky

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3291038

RESULTS

PARTICIPANT FLOW:
Groups:
- Vehicle Ointment: Participants applied vehicle ointment topically twice a day (BID) to the stasis dermatitis affected lower extremities (knees to feet) for 6 weeks. Participants were followed-up for 4 weeks after treatment completion.
- Crisaborole 2% Ointment: Participants applied crisaborole ointment 2 percent (%) topically BID to the stasis dermatitis affected lower extremities (knees to feet) for 6 weeks. Participants were followed-up for 4 weeks after treatment completion.
Period: Overall Study
Arm/Group | Vehicle Ointment | Crisaborole 2% Ointment
Started | 33 | 33
Treated | 32 | 33
Completed | 23 | 26
Not Completed | 10 | 7
Not completed — Not treated | 1 | 0
Not completed — Adverse Event | 4 | 4
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 5 | 2

BASELINE CHARACTERISTICS:
Population: Full analysis set included all participants who were randomly assigned to study intervention and applied at least 1 dose of study intervention. Participants were analyzed according to the intervention they were randomized.
Groups:
- Vehicle Ointment: Participants applied vehicle ointment topically BID to the stasis dermatitis affected lower extremities (knees to feet) for 6 weeks. Participants were followed-up for 4 weeks after treatment completion.
- Crisaborole 2% Ointment: Participants applied crisaborole ointment 2% topically BID to the stasis dermatitis affected lower extremities (knees to feet) for 6 weeks. Participants were followed-up for 4 weeks after treatment completion.
- Total: Total of all reporting groups
Arm/Group | Vehicle Ointment | Crisaborole 2% Ointment | Total
Number analyzed (Participants) | 32 | 33 | 65
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.9 (9.81) | 66.0 (8.64) | 67.4 (9.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 18 | 17 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 31 | 30 | 61
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 31 | 29 | 60
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Total Sign Score (TSS) at Week 6: In-person Assessment
Description: TSS assesses severity of stasis dermatitis lesions. There were following 4 clinical signs of all treatable stasis dermatitis lesions: erythema, papulation/elevation, superficial erosion/denudation, and scaling. Each of 4 signs were rated on a scale of 0 to 3 (0= none, 1= mild, 2= moderate, 3= severe). TSS = sum of scores from all clinical signs; ranging from 0 (none) to 12 (most severe), where higher score indicated greater severity. The assessment was completed in person by the home visit practitioner.
Time Frame: Baseline, Week 6
Population: Full analysis set included all participants who were randomly assigned to study intervention and applied at least 1 dose of study intervention. Participants were analyzed according to the intervention they were randomized. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Vehicle Ointment | Crisaborole 2% Ointment
Number analyzed (Participants) | 26 | 30
Percent change | -18.07 (5.47) | -32.44 (5.09)
Statistical Analysis 1: Comparison: Vehicle Ointment vs Crisaborole 2% Ointment; Test type: Superiority; p = 0.0299, ANOVA — 1-sided; Least square (LS) mean difference = -14.36, 90% CI 2-sided [-26.87 to -1.86], Standard Error of Mean 7.47

2. Secondary Outcome: Percentage of Participants Who Achieved Treatment Success Based on Investigator's Static Global Assessment (ISGA) at Week 6: In-person Assessment
Description: ISGA is a global assessment of stasis dermatitis lesions severity based on erythema, papulation/elevation, superficial erosion/denudation, and scaling. ISGA excludes scalp from scoring and assessment. ISGA score ranged from 0 to 4; where 0 = clear (minor residual hypo/hyperpigmentation; no erythema or induration/papulation; no oozing/crusting), 1= almost clear (trace faint pink erythema, with barely perceptible induration/papulation and no oozing/crusting), 2= mild (faint pink erythema with mild induration/papulation and no oozing/crusting), 3= moderate (pink-red erythema with moderate induration/papulation with or without oozing/crusting), 4= severe (deep or bright red erythema with severe induration/papulation and with oozing/crusting). Higher scores indicated greater severity. The assessment was completed in person by the home visit practitioner. Treatment success was defined as ISGA score of clear/almost clear with at least a 2-grade improvement from baseline.
Time Frame: Week 6
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Vehicle Ointment | Crisaborole 2% Ointment
Number analyzed (Participants) | 26 | 30
Percentage of participants | 0 | 3.33
Statistical Analysis 1: Comparison: Vehicle Ointment vs Crisaborole 2% Ointment; Test type: Superiority; p = 0.1546, Normal approximation test — 1-sided; Difference in percentage of participants = 3.33, 90% CI 2-sided [-2.06 to 8.72]

3. Secondary Outcome: Percentage of Participants Who Achieved Treatment Success Based on Investigator's Static Global Assessment (ISGA) at Week 1, 2, 3, 4, 5 and 6: Central Readers Digital Images Assessment
Description: ISGA: global assessment of stasis dermatitis lesions severity based on erythema, papulation/elevation, superficial erosion/denudation, and scaling, excluding scalp. ISGA score ranged from 0 to 4; 0 = clear (minor residual hypo/hyperpigmentation; no erythema or induration/papulation; no oozing/crusting), 1= almost clear (trace faint pink erythema, with barely perceptible induration/papulation and no oozing/crusting), 2= mild (faint pink erythema with mild induration/papulation and no oozing/crusting), 3= moderate (pink-red erythema with moderate induration/papulation with or without oozing/crusting), 4= severe (deep or bright red erythema with severe induration/papulation and with oozing/crusting). Higher scores = greater severity. Treatment success: ISGA score of clear/almost clear with at least a 2-grade improvement from baseline. Participants acquired static digital images of the lesions using sponsor-provisioned digital imaging equipment. Images were reviewed by central readers.
Time Frame: Week 1, 2, 3, 4, 5 and 6
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Vehicle Ointment | Crisaborole 2% Ointment
Number analyzed (Participants) | 32 | 33
Percentage of participants
  Week 1 | 3.13 | 12.12
  Week 2 | 15.63 | 15.15
  Week 3 | 12.50 | 12.12
  Week 4 | 12.50 | 12.12
  Week 5 | 6.25 | 15.15
  Week 6 | 0 | 18.18
Statistical Analysis 1: Comparison: Vehicle Ointment vs Crisaborole 2% Ointment; Week 1; Test type: Superiority; p = 0.0819, Normal approximation test — 1-sided; Difference in percentage of participants = 9.00, 90% CI 2-sided [-1.63 to 19.62]
Statistical Analysis 2: Comparison: Vehicle Ointment vs Crisaborole 2% Ointment; Week 2; Test type: Superiority; p = 0.4789, Normal approximation test — 1-sided; Difference in percentage of participants = -0.47, 90% CI 2-sided [-15.20 to 14.25]
Statistical Analysis 3: Comparison: Vehicle Ointment vs Crisaborole 2% Ointment; Week 3; Test type: Superiority; p = 0.4815, Normal approximation test — 1-sided; Difference in percentage of participants = -0.38, 90% CI 2-sided [-13.79 to 13.03]
Statistical Analysis 4: Comparison: Vehicle Ointment vs Crisaborole 2% Ointment; Week 4; Test type: Superiority; p = 0.4815, Normal approximation test — 1-sided; Difference in percentage of participants = -0.38, 90% CI 2-sided [-13.79 to 13.03]
Statistical Analysis 5: Comparison: Vehicle Ointment vs Crisaborole 2% Ointment; Week 5; Test type: Superiority; p = 0.1197, Normal approximation test — 1-sided; Difference in percentage of participants = 8.90, 90% CI 2-sided [-3.55 to 21.35]
Statistical Analysis 6: Comparison: Vehicle Ointment vs Crisaborole 2% Ointment; Week 6; Test type: Superiority; p = 0.0034, Normal approximation test — 1-sided; Difference in percentage of participants = 18.18, 90% CI 2-sided [7.14 to 29.23]

4. Secondary Outcome: Percentage of Participants With an Investigator's Static Global Assessment (ISGA) Score of Clear (0) or Almost Clear (1) at Week 6: In-person Assessment
Description: ISGA is a global assessment of stasis dermatitis lesions severity based on erythema, papulation/elevation, superficial erosion/denudation, and scaling. ISGA excludes scalp from scoring and assessment. ISGA score ranged from 0 to 4; where 0 = clear (minor residual hypo/hyperpigmentation; no erythema or induration/papulation; no oozing/crusting), 1= almost clear (trace faint pink erythema, with barely perceptible induration/papulation and no oozing/crusting), 2= mild (faint pink erythema with mild induration/papulation and no oozing/crusting), 3= moderate (pink-red erythema with moderate induration/papulation with or without oozing/crusting), 4= severe (deep or bright red erythema with severe induration/papulation and with oozing/crusting). Higher scores indicated greater severity. The assessment was completed in person by the home visit practitioner.
Time Frame: Week 6
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Vehicle Ointment | Crisaborole 2% Ointment
Number analyzed (Participants) | 26 | 30
Percentage of participants | 11.54 | 16.67
Statistical Analysis 1: Comparison: Vehicle Ointment vs Crisaborole 2% Ointment; Test type: Superiority; p = 0.2896, Normal approximation test — 1-sided; Difference in percentage of participants = 5.13, 90% CI 2-sided [-10.09 to 20.34]

5. Secondary Outcome: Percentage of Participants With an Investigator's Static Global Assessment (ISGA) Score of Clear (0) or Almost Clear (1) at Week 1, 2, 3, 4, 5 and 6: Central Readers Digital Images Assessment
Description: ISGA is a global assessment of stasis dermatitis lesions severity based on erythema, papulation/elevation, superficial erosion/denudation, and scaling. ISGA excludes scalp from scoring and assessment. ISGA score ranged from 0 to 4; where 0 = clear (minor residual hypo/hyperpigmentation; no erythema or induration/papulation; no oozing/crusting), 1= almost clear (trace faint pink erythema, with barely perceptible induration/papulation and no oozing/crusting), 2= mild (faint pink erythema with mild induration/papulation and no oozing/crusting), 3= moderate (pink-red erythema with moderate induration/papulation with or without oozing/crusting), 4= severe (deep or bright red erythema with severe induration/papulation and with oozing/crusting). Higher scores indicated greater severity. Participants acquired static digital images of the lesions using sponsor-provisioned digital imaging equipment. Images were reviewed by central readers.
Time Frame: Week 1, 2, 3, 4, 5 and 6
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Vehicle Ointment | Crisaborole 2% Ointment
Number analyzed (Participants) | 32 | 33
Percentage of participants
  Week 1 | 43.75 | 51.52
  Week 2 | 37.50 | 54.55
  Week 3 | 43.75 | 45.45
  Week 4 | 43.75 | 45.45
  Week 5 | 25.00 | 45.45
  Week 6 | 21.88 | 51.52
Statistical Analysis 1: Comparison: Vehicle Ointment vs Crisaborole 2% Ointment; Week 1; Test type: Superiority; p = 0.2648, Normal approximation test — 1-sided; Difference in percentage of participants = 7.77, 90% CI 2-sided [-12.55 to 28.08]
Statistical Analysis 2: Comparison: Vehicle Ointment vs Crisaborole 2% Ointment; Week 2; Test type: Superiority; p = 0.0809, Normal approximation test — 1-sided; Difference in percentage of participants = 17.05, 90% CI 2-sided [-2.99 to 37.08]
Statistical Analysis 3: Comparison: Vehicle Ointment vs Crisaborole 2% Ointment; Week 3; Test type: Superiority; p = 0.4450, Normal approximation test — 1-sided; Difference in percentage of participants = 1.70, 90% CI 2-sided [-18.58 to 21.99]
Statistical Analysis 4: Comparison: Vehicle Ointment vs Crisaborole 2% Ointment; Week 4; Test type: Superiority; p = 0.4450, Normal approximation test — 1-sided; Difference in percentage of participants = 1.70, 90% CI 2-sided [-18.58 to 21.99]
Statistical Analysis 5: Comparison: Vehicle Ointment vs Crisaborole 2% Ointment; Week 5; Test type: Superiority; p = 0.0385, Normal approximation test — 1-sided; Difference in percentage of participants = 20.45, 90% CI 2-sided [1.43 to 39.48]
Statistical Analysis 6: Comparison: Vehicle Ointment vs Crisaborole 2% Ointment; Week 6; Test type: Superiority; p = 0.0045, Normal approximation test — 1 sided; Difference in percentage of participants = 29.64, 90% CI 2-sided [10.95 to 48.33]

6. Secondary Outcome: Percent Change From Baseline in Total Sign Score (TSS) at Week 1, 2, 3, 4, 5 and 6: Central Readers Digital Images Assessment
Description: TSS assesses severity of stasis dermatitis lesions. There were following 4 clinical signs of all treatable stasis dermatitis lesions: erythema, papulation/elevation, superficial erosion/denudation, and scaling. Each of 4 signs were rated on a scale of 0 to 3 (0= none, 1= mild, 2= moderate, 3= severe). TSS = sum of scores from all clinical signs; ranging from 0 (none) to 12 (most severe), where higher score indicated greater severity. Participants acquired static digital images of the lesions using sponsor-provisioned digital imaging equipment. Images were reviewed by central readers.
Time Frame: Baseline, Week 1, 2, 3, 4, 5 and 6
Population: Full analysis set included all participants who were randomly assigned to study intervention and applied at least 1 dose of study intervention. Participants were analyzed according to the intervention they were randomized. Here, "number analyzed" signifies participants evaluable for the specified rows.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Vehicle Ointment | Crisaborole 2% Ointment
Number analyzed (Participants) | 32 | 33
Percent change
  Week 1: number analyzed (Participants) | 29 | 29
  Week 1 | -20.35 (9.55) | -16.48 (9.52)
  Week 2: number analyzed (Participants) | 27 | 26
  Week 2 | -35.94 (8.14) | -40.41 (8.26)
  Week 3: number analyzed (Participants) | 24 | 26
  Week 3 | -34.86 (10.26) | -25.05 (9.85)
  Week 4: number analyzed (Participants) | 25 | 25
  Week 4 | -39.38 (11.14) | -4.64 (11.12)
  Week 5: number analyzed (Participants) | 22 | 23
  Week 5 | -27.23 (10.41) | -28.89 (10.18)
  Week 6: number analyzed (Participants) | 21 | 22
  Week 6 | -10.29 (8.60) | -52.48 (8.35)
Statistical Analysis 1: Comparison: Vehicle Ointment vs Crisaborole 2% Ointment; Week 1; Test type: Superiority; p = 0.3874, Normal approximation test — 1-sided; LS mean Difference = 3.88, 90% CI 2-sided [-18.67 to 26.43], Standard Error of Mean 13.49
Statistical Analysis 2: Comparison: Vehicle Ointment vs Crisaborole 2% Ointment; Week 2; Test type: Superiority; p = 0.3506, Normal approximation test — 1-sided; LS mean Difference = -4.47, 90% CI 2-sided [-23.85 to 14.91], Standard Error of Mean 11.59
Statistical Analysis 3: Comparison: Vehicle Ointment vs Crisaborole 2% Ointment; Week 3; Test type: Superiority; p = 0.2466, Normal approximation test — 1-sided; LS mean Difference = 9.81, 90% CI 2-sided [-13.97 to 33.60], Standard Error of Mean 14.23
Statistical Analysis 4: Comparison: Vehicle Ointment vs Crisaborole 2% Ointment; Week 4; Test type: Superiority; p = 0.0157, Normal approximation test — 1-sided; LS mean Difference = 34.74, 90% CI 2-sided [8.43 to 61.05], Standard Error of Mean 15.74
Statistical Analysis 5: Comparison: Vehicle Ointment vs Crisaborole 2% Ointment; Week 5; Test type: Superiority; p = 0.4548, Normal approximation test — 1-sided; LS mean Difference = -1.66, 90% CI 2-sided [-25.99 to 22.68], Standard Error of Mean 14.55
Statistical Analysis 6: Comparison: Vehicle Ointment vs Crisaborole 2% Ointment; Week 6; Test type: Superiority; p = 0.0004, Normal approximation test — 1-sided; LS mean Difference = -42.19, 90% CI 2-sided [-62.24 to -22.15], Standard Error of Mean 11.99

7. Secondary Outcome: Percent Change From Baseline in Stasis Dermatitis Lesional Percent Body Surface Area (BSA) at Week 6: In-person Assessment
Description: Stasis dermatitis lesional BSA was calculated using handprint method. Number of handprints (size of participant's full palmer hand) fitting in affected area was counted. One handprint represented approximately 1% of lesional BSA. Percent BSA for a body region = total number of handprints in a body region * % surface area equivalent to 1 handprint. Higher % BSA indicated greater severity. The assessment was completed in person by the home visit practitioner.
Time Frame: Baseline, Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Vehicle Ointment | Crisaborole 2% Ointment
Number analyzed (Participants) | 26 | 30
Percent change | -10.72 (7.06) | -3.80 (6.57)
Statistical Analysis 1: Comparison: Vehicle Ointment vs Crisaborole 2% Ointment; Test type: Superiority; p = 0.2383, ANOVA — 1 sided; LS mean difference = 6.91, 90% CI 2-sided [-9.23 to 23.06], Standard Error of Mean 9.65

8. Secondary Outcome: Percent Change From Baseline in Percent Body Surface Area (BSA) at Week 1, 2, 3, 4, 5 and 6: Central Readers Digital Images Assessment
Description: Stasis dermatitis lesional BSA was calculated using handprint method. Number of handprints (size of participant's full palmer hand) fitting in affected area was counted. One handprint represented approximately 1% of lesional BSA. Percent BSA for a body region = total number of handprints in a body region * % surface area equivalent to 1 handprint. Higher % BSA indicated greater severity. Participants acquired static digital images of the lesions using sponsor-provisioned digital imaging equipment. Images were reviewed by central readers.
Time Frame: Baseline, Week 1, 2, 3, 4, 5 and 6
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Vehicle Ointment | Crisaborole 2% Ointment
Number analyzed (Participants) | 32 | 33
Percent change
  Week 1: number analyzed (Participants) | 29 | 28
  Week 1 | 10.28 (14.73) | -19.67 (14.98)
  Week 2: number analyzed (Participants) | 27 | 25
  Week 2 | -13.21 (13.07) | -27.59 (13.50)
  Week 3: number analyzed (Participants) | 24 | 26
  Week 3 | -31.58 (10.85) | -41.52 (10.44)
  Week 4: number analyzed (Participants) | 25 | 24
  Week 4 | -2.34 (15.80) | -18.35 (15.93)
  Week 5: number analyzed (Participants) | 22 | 22
  Week 5 | -6.05 (13.87) | -19.06 (13.91)
  Week 6: number analyzed (Participants) | 21 | 21
  Week 6 | 18.67 (21.26) | -34.34 (21.23)
Statistical Analysis 1: Comparison: Vehicle Ointment vs Crisaborole 2% Ointment; Week 1; Test type: Superiority; p = 0.0797, Normal approximation test — 1-sided; LS mean Difference = -29.95, 90% CI 2-sided [-65.09 to 5.18], Standard Error of Mean 21.01
Statistical Analysis 2: Comparison: Vehicle Ointment vs Crisaborole 2% Ointment; Week 2; Test type: Superiority; p = 0.2236, Normal approximation test — 1-sided; LS mean Difference = -14.39, 90% CI 2-sided [-45.81 to 17.04], Standard Error of Mean 18.79
Statistical Analysis 3: Comparison: Vehicle Ointment vs Crisaborole 2% Ointment; Week 3; Test type: Superiority; p = 0.2559, Normal approximation test — 1-sided; LS mean Difference = -9.94, 90% CI 2-sided [-35.12 to 15.24], Standard Error of Mean 15.05
Statistical Analysis 4: Comparison: Vehicle Ointment vs Crisaborole 2% Ointment; Week 4; Test type: Superiority; p = 0.2392, Normal approximation test — 1-sided; LS mean Difference = -16.01, 90% CI 2-sided [-53.54 to 21.52], Standard Error of Mean 22.44
Statistical Analysis 5: Comparison: Vehicle Ointment vs Crisaborole 2% Ointment; Week 5; Test type: Superiority; p = 0.2553, Normal approximation test — 1-sided; LS mean Difference = -13.01, 90% CI 2-sided [-45.87 to 19.85], Standard Error of Mean 19.65
Statistical Analysis 6: Comparison: Vehicle Ointment vs Crisaborole 2% Ointment; Week 6; Test type: Superiority; p = 0.0416, Normal approximation test — 1-sided; LS mean Difference = -53.01, 90% CI 2-sided [-103.26 to -2.75], Standard Error of Mean 30.05

9. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) was any untoward medical occurrence attributed to a participant who received study drug without regard to possibility of causal relationship. Treatment-emergent were events between first dose of study drug and up to 4 weeks after last dose that were absent before treatment or that worsened relative to pre-treatment state. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; Initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. TEAEs included both SAEs and all non-SAEs.
Time Frame: Day 1 up to maximum of 4 weeks after the last dose (maximum for 10 weeks)
Population: Safety analysis set included all participants who were randomly assigned to study intervention and applied at least 1 dose of study intervention and were analyzed according to intervention actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle Ointment | Crisaborole 2% Ointment
Number analyzed (Participants) | 32 | 33
Participants
  TEAEs | 14 | 13
  SAEs | 4 | 1

ADVERSE EVENTS:
Time Frame: Day 1 up to maximum of 4 weeks after the last dose (maximum for 10 weeks)
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Safety analysis set included all participants who were randomly assigned to study intervention and applied at least 1 dose of study intervention and were analyzed according to intervention actually received.
Arm/Group | Vehicle Ointment | Crisaborole 2% Ointment
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/33
Serious Adverse Events (participants affected / at risk) | 4/32 | 1/33
Other Adverse Events (participants affected / at risk) | 13/32 | 13/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vehicle Ointment (N=32) | Crisaborole 2% Ointment (N=33)
Muscular dystrophy (Congenital, familial and genetic disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1
Cystitis (Infections and infestations) | 1 | 0
Oropharyngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vehicle Ointment (N=32) | Crisaborole 2% Ointment (N=33)
Muscular dystrophy (Congenital, familial and genetic disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Oesophageal spasm (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Injection site erythema (General disorders) | 0 | 1
Injection site pruritus (General disorders) | 0 | 1
Oedema (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Peripheral swelling (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 1
Bronchitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Conjunctivitis viral (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Tinea pedis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 2
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Burning sensation (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 2
Migraine (Nervous system disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 2
Erythema (Skin and subcutaneous tissue disorders) | 2 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3
Skin erosion (Skin and subcutaneous tissue disorders) | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0
Hot flush (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-07-19): https://cdn.clinicaltrials.gov/large-docs/87/NCT04091087/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-16): https://cdn.clinicaltrials.gov/large-docs/87/NCT04091087/SAP_001.pdf